CLINICAL TRIAL: NCT02117167
Title: Intergroup Trial UNICANCER UC 0105-1305/ IFCT 1301: SAFIR02_Lung - Evaluation of the Efficacy of High Throughput Genome Analysis as a Therapeutic Decision Tool for Patients With Metastatic Non-small Cell Lung Cancer
Brief Title: SAFIR02_Lung - Efficacy of Targeted Drugs Guided by Genomic Profiles in Metastatic NSCLC Patients
Acronym: SAFIR02_Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Intergroupe Francophone de Cancerologie Thoracique (Other); Fondation ARC (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0105/1305 / IFCT 1301; 2013-001653-27 (EudraCT Number)
Record Dates: First submitted 2014-04-08; First posted 2014-04-17 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Non-small Cell Lung Cancer Metastatic
MeSH Terms: interventions — vistusertib; AZD4547; capivasertib; AZD 8931; AZD 6244; vandetanib; Pemetrexed; durvalumab; 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Substudy 1: targeted agent (Experimental): Arm A1/ targeted arm: targeted maintenance from a list of targeted drugs guided by the genomic analysis, AZD2014 tablet per os 50 mg bd, continuous dosing, AZD4547 tablet per os 80 mg bd, 2 weeks on/1 week off, AZD5363 capsule per os 480 mg bd, 4 days on/3 days off, AZD8931 tablet per os 40 mg bd, continuous dosing, selumetinib capsule per os 75 mg bd, continuous dosing, vandetanib tablet per os 300 mg od, continuous dosing, olaparib tablet per os 300 mg bd continuous dosing savolitinib tablet per os 600 mg od continuous dosing
  Interventions: Drug: AZD2014; Drug: AZD4547; Drug: AZD5363; Drug: AZD8931; Drug: Selumetinib; Drug: Vandetanib; Drug: savolitinib; Drug: Olaparib
- Substudy 1: standard maintenance therapy (Active Comparator): Arm B1/ standard arm pemetrexed Intra venous 500 mg/m², every 3 weeks, standard maintenance left to the investigator's choice
  Interventions: Drug: Standard maintenance for squamous NSCLC; Drug: Pemetrexed
- Substudy 2: Immunotherapy (Experimental): Arm A2/ Immunotherapy arm: maintenance with durvalumab for patient without actionable genomic alterations or non eligible to Targeted substudy 1, durvalumab Intra-venous 10 mg/kg, Q2W
  Interventions: Drug: Durvalumab
- Substudy 2: standard maintenance therapy (Active Comparator): Arm B2/ standard arm pemetrexed Intra venous 500 mg/m², every 3 weeks, standard maintenance left to the investigator's choice
  Interventions: Drug: Standard maintenance for squamous NSCLC; Drug: Pemetrexed

INTERVENTIONS:
Drug: AZD2014 — Target: m-TOR
  Arms: Substudy 1: targeted agent
Drug: AZD4547 — Target: FGFR
  Arms: Substudy 1: targeted agent
Drug: AZD5363 — Target: AKT
  Arms: Substudy 1: targeted agent
Drug: AZD8931 — Target: HER2, EGFR
  Arms: Substudy 1: targeted agent
Drug: Selumetinib — Target: MEK
  Other Names: ARRY-142866
  Arms: Substudy 1: targeted agent
Drug: Vandetanib — Target : VEGF, EGFR
  Other Names: CAPRELSA
  Arms: Substudy 1: targeted agent
Drug: Standard maintenance for squamous NSCLC
  Arms: Substudy 1: standard maintenance therapy; Substudy 2: standard maintenance therapy
Drug: Pemetrexed — Standard maintenance for non squamous NSCLC
  Other Names: ALIMTA
  Arms: Substudy 1: standard maintenance therapy; Substudy 2: standard maintenance therapy
Drug: Durvalumab — Target: PD-L1
  Arms: Substudy 2: Immunotherapy
Drug: savolitinib — target : MET
  Arms: Substudy 1: targeted agent
Drug: Olaparib — target : PARP
  Other Names: LYNPARZA
  Arms: Substudy 1: targeted agent

SUMMARY:
Open label multicentric randomized phase II trial, using high throughput genome analysis as a therapeutic decision tool, aimed at comparing a targeted treatment administered according to the identified molecular anomalies of the tumor with a standard treatment (pemetrexed in Non-squamous patients and erlotinib in squamous cells, targeted substudy 1) as well as immunotherapy with maintenance therapy in patients without actionable genomic alterations or non eligible to substudy 1 (immune substudy 2).

DETAILED DESCRIPTION:
Screening phase:

New frozen biopsy or an archived frozen sample or ctDNA sample will be sent to the genomic platforms for DNA extraction and genomic analysis (DNA microarrays and Next generation sequencing).

Patients can be considered as pre-eligible for the targeted substudy 1 randomisation phase when both following mandatory conditions have been met : stable or responding disease has been observed after 4 cycles of chemotherapy (investigator judgment) and targetable alteration has been identified by the Molecular tumor board (MTB).

If not eligible for the substudy 1 randomisation phase, patients can be considered as pre-eligible for the immune substudy 2 randomization phase when both following mandatory conditions are met: stable or responding disease (investigator judgment) is observed after 4 cycles of a platinum-based chemotherapy AND not eligible to randomization in the substudy 1 (because patient had no targetable alteration identified by the Molecular Tumor Board, or failed to have a genomic profile for the tumor [low tumor cells percentage, technical issue during genomic analysis, etc.], or a non-inclusion criteria that precluded entry into the substudy 1)

Randomization phase:

The mandatory post-chemotherapy 28-day wash-out period following cycle 4 of chemotherapy will provide time to achieve all the required tests and examinations.

The randomization program will allocate the following treatments with a 2:1 ratio in favor of Arm A of the considered substudy:

Substudy 1 : targeted therapies versus standard maintenance therapy

* Arm A1 / targeted arm: targeted maintenance from a list of 6 targeted drugs guided by the genomic analysis, or
* Arm B1 / standard arm : standard maintenance (pemetrexed in non-squamous and standard practice in squamous NSCLC).

Substudy 2 : immunotherapy versus standard maintenance therapy

* Arm A2 / immunotherapy maintenance arm: MEDI4736 or
* Arm B2 / standard arm : standard maintenance (pemetrexed in non-squamous and standard practice in squamous NSCLC).

ELIGIBILITY:
Screening phase:

Inclusion Criteria:

* histologically proven NSCLC
* Metastatic relapse or stage IV at diagnosis, or stage IIIb not amenable to surgery or radiotherapy
* No EGFR-activating mutation or ALK translocation
* primary tumor or metastases that can be biopsied, excluding bone.
* Age >18 years
* WHO Performance Status 0/1
* Chemo-naïve patients eligible to a first line platinum-based chemotherapy
* No tumor progression observed with the current line of treatment
* measurable target lesion or evaluable diseases RECIST

Exclusion criteria

* Spinal cord compression and/or symptomatic or progressive brain metastases
* Abnormal coagulation contraindicating biopsy
* Inability to swallow
* Major problem with intestinal absorption
* Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG
* Any factors increasing the risk of QTc prolongation or arrhythmic events
* Experience of any of the following in the preceding 12 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, past or current uncontrolled angina pectoris, congestive heart failure NYHA Grade ≥2, torsades de pointes, current uncontrolled hypertension, cardiomyopathy
* Past medical history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which requires steroid treatment or any evidence of clinically interstitial lung disease
* Previous or current malignancies of other histologies within the last 5 years,
* Evidence of severe or uncontrolled systemic disease (active bleeding diatheses, or active Hepatitis B, C and HIV)
* Diagnosis of diabetes mellitus type I or II
* diagnosis of acne rosacea, severe psoriasis and severe atopic eczema
* Prior exposure to anthracyclines or mitoxantrone with cumulative exposure in excess of 360 mg/m² for doxorubicin, 720 mg/m² for epirubicin, or 72 mg/m² for mitoxantrone
* History of retinal degenerative disease, eye injury or corneal surgery in the previous 3 months, past history of central serous retinopathy or retinal vein occlusion, intraocular pressure >21 mmHg, or uncontrolled glaucoma.
* History of hemorrhagic or thrombotic stroke, TIA or other CNS bleeds
* Renal disease including glomerulonephritis, nephritic syndrome, Fanconi syndrome, renal tubular acidosis
* Patients using drugs that are known potent inhibitors or potent inducers or substrates of cytochrome P450

Randomized phase:

Substudy 1:

Inclusion criteria

* Patients who received 4 cycles of an induction platinum-based chemotherapy and who have a SD or a PR at randomization
* presenting at least one genomic alteration from the predefined list
* Age > 25 years for patients planned to receive AZD4547
* 28-day washout period from chemo prior to randomization and grade ≤1 residual toxicities

Exclusion criteria

* Life expectancy <3 months
* Disease progression occuring at any time during chemotherapy and before randomization or toxicity that led to the discontinuation of the platinum-based chemotherapy before 4 full cycles have been delivered
* Less than 28 days from radiotherapy, less than 2 weeks from palliative radiation
* Patients previously treated with a targeted agent in the same class as agents tested in this study
* Toxicities of grade ≥2 from any previous anti-cancer therapy
* Altered haematopoietic or organ function
* Mean resting corrected QT interval (QTc) >480msec (or QTcF >450 msec) obtained from 3 consecutive ECGs
* Left ventricular ejection fraction (LVEF) <55% (MUGA scan or Echocardiogram),
* Altered ophthalmic conditions confirmed by an ophthalmology specialist for patients likely to be treated with AZD4547 orAZD8931 or Selumetinib
* Patients using non-substitutable drugs, that are known to prolong QT interval or induce Torsades de Pointes, when they are supposed to be treated with vandetanib, AZD5363 or AZD8931

Substudy 2:

Inclusion criteria

* Patients who received 4 cycles of an induction platinum-based chemotherapy and who have a SD or a PR at randomization
* Patients not eligible to substudy 1
* 28-day washout period from chemo prior to randomization and grade ≤1 residual toxicities

Exclusion criteria

* Life expectancy <3 months
* Disease progression occuring at any time during chemotherapy and before randomization or toxicity that led to the discontinuation of the platinum-based chemotherapy before 4 full cycles have been delivered
* Any previous treatment with a PD1 or PD-L1 inhibitor, including MEDI4736
* Toxicities of grade ≥2 from any previous anti-cancer therapy
* Altered haematopoietic or organ function
* Mean resting QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 consecutive ECGs using Bazett's Correction
* Current or prior use of immunosuppressive medication within 28 days before the first dose of MEDI4736, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
* History of primary immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 999 (Actual)
Dates: Start 2014-04-23 (Actual); Primary Completion 2018-12-22 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
progression-free survival in the targeted drug arm compared to standard maintenance therapy arm | from randomization to disease progression or death from any cause, whichever comes first, up to 16 months (estimated treatment duration average: 4 months)
  To evaluate whether treatment with targeted agents guided by high throughput molecular analysis (CGH array, next generation sequencing) improves progression-free survival as compared to standard maintenance therapy in patients with metastatic NSCLC

SECONDARY OUTCOMES:
progression-free survival in patients treated with anti-PDL1 antibody (MEDI4736) compared to standard maintenance therapy arm | from randomization to disease progression or death from any cause, whichever comes first, up to 16 months (estimated treatment duration average: 4 months)
  To evaluate whether treatment with MEDI4736 improves progression-free survival as compared to standard maintenance therapy in patients with metastatic NSCLC
overall survival in each substudy | from randomization to death (any cause), up to 16 months
  To evaluate whether treatment with targeted agents guided by high throughput molecular analysis (CGH array, next generation sequencing) or MEDI4736 improves overall survival as compared to standard maintenance therapy in patients with metastatic NSCLC
overall response rates and changes in tumor size in each substudy | tumor response is assessed every 21 days from treatment initiation until first progression or death from any cause, whichever comes first, up to 16 months (estimated treatment duration average: 4 months)
  tumor response is defined as a complete or partial response, upon RECIST v1.1 criteria
evaluate safety, in each substudy | toxicities will be assessed during the whole treatment period (4 months expected in average) followed by a 1-year post-treatment follow-up period, and reported during the visits scheduled by the study flow chart
  Toxicities are graded according to the CTCAE V4
efficacy (response rate, change in tumor size, progression-free survival, overall survival) and safety of each individual targeted agent (substudy 1) | tumor response is assessed every 21 days from treatment initiation until first progression or death from any cause, whichever comes first, up to 16 months (estimated treatment duration average: 4 months)
  tumor response is defined as a complete or partial response, upon RECIST v1.1 criteria
correlate molecular characteristics in patients with the efficacy endpoints (response rate, progression-free and overall survival) in each substudy | from randomization or treatment initiation to disease progression or death from any cause, whichever comes first, up to 16 months (estimated treatment duration average: 4 months)
  tumor response is defined as a complete or partial response, upon RECIST v1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice BARLESI, Pr, Principal Investigator — CHU Hopital Nord Marseille
Locations (37):
- France (37):
  - Centre Hospitalier Henri Duffau, Avignon
  - Centre Hospitalier Universitaire de Besancon - Hopital Jean Minjoz, Besançon
  - Hôpital Avicenne, Bobigny
  - Institut Bergonié, Bordeaux
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Hospices Civils de Lyon- Hôpital Louis Pradel, Bron
  - Centre François Baclesse, Caen
  - CHU Caen, Caen
  - Chu de Caen - Hopital Cote de Nacre, Caen
  - Hôpital Louis Pasteur, Chartres
  - centre Jean Perrin, Clermont-Ferrand
  - CHU Clermont Ferrand - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hopitaux Civils de Colmar, Colmar
  - Centre Hopsitalier Intercommunal de Créteil, Créteil
  - Centre Georges François Leclerc, Dijon
  - CHU Grenoble, Grenoble
  - Chd Vendee, La Roche-sur-Yon
  - CH du Mans, Le Mans
  - Centre Oscar Lambret, Lille
  - CHRU de Lille, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Nord, Marseille
  - Institut Paoli Calmettes, Marseille
  - Institut de cancérologie de l'Ouest, Nantes
  - Centre Antoine Lacassagne, Nice
  - Chr Orleans, Orléans
  - AH-HP Hôpital Saint Louis, Paris
  - AP-HP Hôpital Cochin, Paris
  - AP-HP Hôpital Tenon, Paris
  - Institut Curie, Paris
  - Centre Hospitalier de Pau, Pau
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Chru Strasbourg - Nouvel Hopital Civil, Strasbourg
  - CHI de Toulon - Hôpital Sainte-Musse, Toulon
  - CHU Toulouse -Hôpital Larrey, Toulouse
  - Hôpital Bretonneau, Tours
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Middleton G, Crack LR, Popat S, Swanton C, Hollingsworth SJ, Buller R, Walker I, Carr TH, Wherton D, Billingham LJ. The National Lung Matrix Trial: translating the biology of stratification in advanced non-small-cell lung cancer. Ann Oncol. 2015 Dec;26(12):2464-9. doi: 10.1093/annonc/mdv394. Epub 2015 Sep 25. PMID 26410619
- See also: Unicancer official website — http://www.unicancer.fr
- See also: Intergroupe Francophone de Cancérologie Thoracique (IFCT) official website — http://www.ifct.fr
- See also: SAFIR01 study results — http://www.ncbi.nlm.nih.gov/pubmed/24508104